CLINICAL TRIAL: NCT06464341
Title: Nodal Burden and Nodal Recurrence in Patients With Isolated Tumor Cells After Neoadjuvant Chemotherapy Treated With Axillary Dissection or Nodal Radiation: the OPBC-05/EUBREAST-14R/ICARO Study
Acronym: ICARO
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00418: bb23Weber
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Axillary lymph node dissection; Isolated tumor cells; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with clinical T1-4 N0-3 breast cancer at diagnosis treated with NAC: This cohort study retrospectively analyzed data from 62 centers in 18 countries, mostly members of the Oncoplastic Breast Consortium (OPBC) network. Patients with clinical T1-4 N0-3 breast cancer at diagnosis treated with neoadjuvant chemotherapy between March 2008 and May 2022 were included if they had isolated tumor cells only. ITCs were defined as clusters of tumor cells ≤0.2 mm or clusters of <200 cells in a single cross-sectional image, determined by sentinel lymph node biopsy, targeted axillary dissection, or the MARI procedure (marking axillary lymph nodes with radioactive iodine seeds). Excluded: patients with inflammatory breast cancer, stage IV disease at presentation, axillary lymph node dissection as a primary procedure, and neoadjuvant endocrine therapy. Also excluded cases with micrometastases or macrometastases in any sentinel lymph nodes at frozen section or final pathology, and those where ITCs were detected by One Step Nucleic Acid Amplification.
  Interventions: Other: Observational study no intervention

INTERVENTIONS:
Other: Observational study no intervention — Observational study no intervention

SUMMARY:
The purposes of this multicenter retrospective cohort study are to determine the residual nodal burden in patients with isolated tumor cells detected in the SLN or the clipped node after NAC and to determine oncologic outcomes in this group of patients after ALND or nodal RT or observation.

DETAILED DESCRIPTION:
In the context of upfront surgery, the extent of disease in the sentinel lymph nodes (SLNs) significantly predicts the chances of additional non-SLN metastases during axillary lymph node dissection (ALND). For patients with minimal SLN disease (isolated tumor cells [ITCs] and micrometastases), the probability of further non-SLN metastases is between 10-20%. In contrast, for patients with macrometastases, the risk increases to 27-33%.

In patients undergoing neoadjuvant chemotherapy (NAC), those with positive SLNs exhibit a greater residual nodal burden compared to those treated with upfront surgery. For patients with remaining micro- or macrometastases post-NAC, additional positive lymph nodes are found in over 60% of ALND specimens, regardless of receptor subtype. Consequently, ALND remains the standard care for any residual nodal disease after NAC.

Residual ITCs after NAC are present in about 1.5% of all patients undergoing NAC. There is limited data on the likelihood of discovering additional positive lymph nodes in this group, with fewer than 35 documented cases examining residual nodal burden. Therefore, the benefit of ALND for minimal residual disease is uncertain, and axillary management for patients with nodal ITCs is not standardized. Although omitting ALND reduces arm morbidity, identifying residual nodal disease can influence adjuvant therapy recommendations. Despite the lack of consensus on the oncologic safety of omitting ALND in this group, care patterns indicate a growing adoption of this approach. Given the rarity of this clinical scenario and the absence of forthcoming prospective studies, this study utilized real-world data from a large international cohort to determine the incidence of residual non-SLN involvement in patients with ITCs in the SLNs post-NAC, and to compare clinical outcomes in patients with and without ALND as definitive axillary treatment.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients affected with T1-4 N0-3 breast cancer
* For cN+: Biopsy proven confirmation is required
* For cN0: any axillary staging technique including palpation is allowed
* Residual ITCs in the SLN or clipped node
* At least 1-year follow-up (12/2021 or later depending on the time of data collection)
* For cN0: SLNB with single or dual tracer mapping
* For cN+: SLNB with dual mapping or targeted axillary dissection (TAD: imaging-guided localization of sampled node in combination with SLN procedure with or without dual mapping)
* Underwent TAD/SLNB +/- ALND +/- axillary RT

Exclusion Criteria:

* Male patients
* Patients with nodal pCR
* Patients with residual nodal micro- or macrometastases
* Stage IV disease at presentation
* Inflammatory breast cancer (T4d) at presentation

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients will be included. There is no formal sample size calculation
Sampling Method: Non-Probability Sample
Enrollment: 583 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Axillary Lymph Node Dissection (ALND) | Day 0
  Evaluation of the number of ALNDs performed
Number of Tailored Axillary Dissection (TAD) | Day 0
  Evaluation of the number of TAD performed
Number of Sentinel Lymph Node Biopsy (SLNB) | one time assessment before surgery
  Evaluation of the number of SLNB performed
Number Axillary Radiotherapy | Up to 2 years
  Evaluation of the number of axillary radiotherapy performed
Number of additional micrometastases | Day 0
  Evaluation of the number of additional micrometastases removed by ALND
Number of additional macrometastases | Day 0
  Evaluation of the number of additional macrometastases removed by ALND
Axillary recurrence | Up to 14 years
  Evaluation of the number of axillary recurrence

SECONDARY OUTCOMES:
Regional recurrence | Up to 14 years
  Evaluation of the number of regional recurrence
Locoregional recurrence | Up to 14 years
  Evaluation of the number of locoregional recurrence
Invasive recurrence | Up to 14 years
  Evaluation of the number of invasive recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Walter P. Weber, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (62):
- United States (20):
  - Valleywise Health Medical Center, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Samuel Oschin Cancer Institute, Los Angeles, California
  - Miami University, Miami, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Guthrie Clinic, Sayre, Pennsylvania
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington, Seattle, Washington
- Medical University of Vienna, Vienna, Austria
- University Hospital Ghent, Ghent, Belgium
- Brazil (5):
  - Sirio-Libanes Hospital, Department of Oncology, Brasília
  - Nossa Senhora das Gracias Hospital, Curitiba
  - Instituto de Mastologia e Oncologia, Goiânia
  - Santa Paula Hospital, São Paulo
  - Sirio-Libanes Hospital, Department of Oncology, São Paulo
- Mc Gill University, Montreal, Canada
- Germany (6):
  - Universitätsklinikum Augsburg, Augsburg
  - University Hospital Düsseldorf, Düsseldorf
  - KEM Evang. Kliniken Essen-Mitte, Essen
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Schleswig-Holstein Campus Lübeck, Lübeck
  - German Breast Group, Neu-Isenburg
- Greece (2):
  - Athens Medical Center, Athens
  - Heraklion University Hospital, Heraklion
- Sheba Medical Center, Tel Litwinsky, Israel
- Italy (5):
  - Instituto Nazionale Tumori (IRCCS), Naples
  - University of Naples Federico, Naples
  - Veneto Institute of Oncology IRCCS, Padua
  - Istituti Clinici Scientifici Maugeri IRCCS,, Pavia
  - IRCCS Humanitas Research Hospital, Rozzano
- Antoni van Leeuwenhoek, Amsterdam, Netherlands
- University Hospital of Zielona Góra, Zielona Góra, Poland
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Korea (3):
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Hospital del Mar, Barcelona, Spain
- Sahlgrenska University Hospital Gothenburg, Gothenburg, Sweden
- Switzerland (4):
  - University Hospital Basel, Basel, Canton of Basel-City
  - Kantonsspital Baden, Baden
  - Breastcenter Zürich, Zurich
  - University Hospital Zürich, Zurich
- Turkey (Türkiye) (6):
  - Gülhane Research and Training Hospital, Ankara
  - Acıbadem Research Instıtute of Senology, Istanbul
  - Istanbul University Institute of Oncology, Istanbul
  - Istanbul University, Faculty of Medicine, Istanbul
  - Marmara University, School of Medicine, Istanbul
  - Zonguldak Bulent Ecevit University, Zonguldak
- United Kingdom (2):
  - Cambridge University Hospital, Cambridge
  - The Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montagna G, Laws A, Ferrucci M, Mrdutt MM, Sun SX, Bademler S, Balbaloglu H, Balint-Lahat N, Banys-Paluchowski M, Barrio AV, Benson J, Bese N, Boughey JC, Boyle MK, Diego EJ, Eden C, Eller R, Goldschmidt M, Hlavin C, Heidinger M, Jelinska J, Karadeniz Cakmak G, Kesmodel SB, King TA, Kuerer HM, Loesch J, Milardi F, Murawa D, Moo TA, Menes TS, Passeri D, Pastoriza JM, Perhavec A, Pislar N, Polidorio N, Rami A, Ryu JM, Schulz A, Sevilimedu V, Ugurlu MU, Uras C, van Hemert A, Wong SM, Yoo TR, Zhang JQ, Karanlik H, Cabioglu N, Peeters MV, Morrow M, Weber WP; ICARO Study Group. Nodal Burden and Oncologic Outcomes in Patients With Residual Isolated Tumor Cells After Neoadjuvant Chemotherapy (ypN0i+): The OPBC-05/ICARO Study. J Clin Oncol. 2025 Mar;43(7):810-820. doi: 10.1200/JCO.24.01052. Epub 2024 Nov 7. PMID 39509672